CLINICAL TRIAL: NCT01093118
Title: A Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of TMI-358 in the Treatment of Distal Subungual Onychomycosis of the Toenail
Brief Title: A Study to Evaluate TMI-358 in the Treatment of Distal Subungual Onychomycosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Talima Therapeutics, Inc. (Industry)
Responsible Party: Martin Babler, Talima Therapeutics, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCP-TMI-7007
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2011-01

CONDITIONS: Distal Subungual Onychomycosis
Keywords: Distal subungual onychomycosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TMI-358 (Experimental): Active treatment
  Interventions: Drug: TMI-358
- MMI-467 (Placebo Comparator)
  Interventions: Drug: MMI-467

INTERVENTIONS:
Drug: TMI-358 — Micro implant monthly x 3
  Arms: TMI-358
Drug: MMI-467 — Micro implant monthly x 3
  Arms: MMI-467

SUMMARY:
The purpose of this study is to determine if a local treatment is effective for the treatment of toenail fungus (distal subungual onychomycosis).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 75 years of age, inclusive
* Diagnosed with distal subungual onychomycosis (DSO) of the toenails
* Great toe(s) with intact skin and intact neurologic functions
* Great toenail(s) free of nail polish
* At least one target great toe which has:

  * 25 to 75% involvement of the area of the nail unit (including destroyed or missing parts of the nail plate)
  * at least 2 mm of uninvolved nail growth as measured from the proximal nail fold to the most proximal point to the disease process and with no lunular involvement
  * nail unit hyperkeratosis at the most distal edge which measures no greater than 3 mm
  * a positive KOH and culture

Exclusion Criteria:

* Any significant disease of the hepatic, renal, endocrine (including diabetes mellitus), immune systems, or other health conditions which could interfere with or confound the results of study assessments
* Pre-existing chronic foot pain, neurologic deficit or skin disease/injury in treated foot
* In the case of female subjects, are pregnant, nursing, or planning to become pregnant within the study period
* History of clinically significant abnormal laboratory values, including liver function test results equal to or greater than 2 x the upper limit of normal
* Disease-like psoriatic toenails, significant toenail abnormalities/dystrophies, toenail injuries or any other condition in the toenail which could interfere with study evaluations (e.g., prevent obtaining normal appearing nail, after clearing of onychomycosis, due to chemical damage, genetic or pigmentary disorders, etc.)
* Have white superficial onychomycosis, proximal subungual onychomycosis, yellow spikes, or dermatophytoma
* Have paronychia
* Have a history of chronic alcohol or drug abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Cure rates | 48 weeks
  Based on clinical evaluations (nail measurements, KOH, and mycological culture for dermatophytes), cure categories will be defined as either mycological cure, clinical cure, complete cure, or effective treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Terry Jones, MD, Principal Investigator — J&S Studies, Inc.; Michael Noss, MD, Principal Investigator — Radiant Research, Inc.; Robert Matheson, MD, Principal Investigator — Oregon Medical Research Center; Leonard Swinyer, MD, Principal Investigator — Dermatology Research Center; Stacy Smith, MD, Principal Investigator — Therapeutics Clinical Research; Norman Bystol, MD, Principal Investigator — Radiant Research, Inc.; Jose Mendez, DO, Principal Investigator — International Dermatology Research Center
Locations (7):
- United States (7):
  - Radiant Research, Inc., Tucson, Arizona
  - Therapeutics Clinical Research, San Diego, California
  - International Dermatology Research Center, Miami, Florida
  - Radiant Research, Inc., Cincinnati, Ohio
  - Oregon Medical Research Center, Portland, Oregon
  - J&S Studies, Inc., College Station, Texas
  - Dermatology Research Center, Salt Lake City, Utah